CLINICAL TRIAL: NCT02243007
Title: Phase II Study of Preoperative FOLFIRINOX Versus Gemcitabine/Nab-Paclitaxel in Patients With Resectable Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David Patrick Ryan, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-218
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Resectable Pancreatic Cancer; Pancreatic Ductal Carcinoma
Keywords: Resectable pancreatic cancer; Pancreatic Ductal Carcinoma
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal | interventions — folfirinox; Radiotherapy; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Folfirinox-ARM A (Experimental): Upon registration patients will be randomized to Arm A (FOLFIRINOX) or Arm B (Gemcitabine/nab-Paclitaxel
  * Treatment will be administered on an outpatient basis and will include intravenous administration of the FOLFIRINOX regimen on predetermined days.
  * After completion of FOLFIRINOX all patients without progressive disease will proceed with radiation therapy with the standard dose of capecitabine.
  * Between 2 and 4 weeks after radiation is complete, patients will proceed for surgical resection of pancreatic cancer
  Interventions: Drug: FOLFIRINOX; Radiation: Radiation therapy; Drug: Capecitabine
- Gemcitabine/nab-Paclitaxel- Arm B (Experimental): * Treatment will be administered on an outpatient basis. Upon registration patients will be randomized to Arm A (FOLFIRINOX) or Arm B (Gemcitabine/nab-Paclitaxel).
  * Intravenous administration of the Gemcitabine/Nab-paclitaxel regimen on predetermined days of each 28 day treatment cycle (unless a delay is mandated by toxicity criteria). A cycle of Gemcitabine/Nab-paclitaxel will constitute a 28 day treatment period.
  * After Gemcitabine/Nab-paclitaxel, all patients without progressive disease will proceed to radiation therapy with the standard dose of capecitabine
  * Between 2 and 4 weeks after radiation is complete, patients will proceed for surgical resection of pancreatic cancer
  Interventions: Drug: Gemcitabine/nab-Paclitaxel; Radiation: Radiation therapy; Drug: Capecitabine

INTERVENTIONS:
Drug: FOLFIRINOX
  Arms: Folfirinox-ARM A
Drug: Gemcitabine/nab-Paclitaxel
  Arms: Gemcitabine/nab-Paclitaxel- Arm B
Radiation: Radiation therapy
Drug: Capecitabine
  Other Names: Xeloda

SUMMARY:
This research study is a Phase II clinical trial, which evaluates a combination of drugs, FOLFIRINOX and Gemcitabine/Nab-Paclitaxel, in the management of participants with resectable pancreatic cancer prior to surgery.

DETAILED DESCRIPTION:
Patients who fulfill eligibility criteria will be randomized to Arm A or Arm B

* Treatment will be administered on an outpatient basis.
* Upon registration participants will be randomized to Arm A (FOLFIRINOX) or Arm B (Gemcitabine/nab-Paclitaxel).
* After completion of FOLFIRINOX or Gemcitabine/Nab-paclitaxel, all participants without progressive disease will proceed to radiation therapy with capecitabine .
* Between 2 and 4 weeks after radiation is complete, participants will proceed for surgical resection of pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

* Cytologic or histologic proof of pancreatic ductal carcinoma is required prior to study entry.
* No evidence of metastatic disease as determined by chest CT scan, and abdominal CT scan (or MRI with gadolinium and/or manganese) and laparoscopy. All patients must be staged with a physical exam, chest CT, abdominal CT with intravenous contrast (or abdominal MRI with gadolinium and/or manganese). Only potentially resectable patients are eligible. Potentially resectable is defined as a) no extrapancreatic disease, b) no evidence (on CT) of involvement of the celiac axis or SMA, c) no evidence (CT or MRI) of occlusion of the SMV or SMPV confluence, and d) no evidence of gross peritoneal or distant metastases by laparoscopy.
* Patients must be 18 years old or older. There will be no upper age restriction.
* ECOG Performance Status of 0 or 1 are eligible.
* Life expectancy of greater than 3 months.
* Lab Values:

  * ANC ≥ 1500 cells/mm3
  * Platelet count at least 100,000 cells/mm3.
  * AST and ALT ≤2.5 x upper limit of normal
  * Total Bilirubin ≤ 5 x upper limit of normal if patient is s/p biliary stenting AND decreasing at least two time points after stenting.
  * Total Bilirubin ≤ 1.5 x upper limit of normal if no biliary stenting was done
  * Serum Creatinine ≤1.5mg/dl OR
  * Creatinine Clearance greater than or equal to 30ml/min (as estimated by Cockroft Gault Equation) (140 - age [yrs]) (body wt [kg])

    * Creatinine clearance for males = ------------ (72) (serum creatinine [mg/dL])
    * Creatinine clearance for females = 0.85 x male value
* The effects of radiation on the developing human fetus are known to be teratogenic. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study treatment plus 30 days from the last date of study drug administration. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Patients who fulfill any of the following criteria will be excluded:

* The presence of metastatic disease on imaging or laparoscopy.
* Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator), such as significant cardiac or pulmonary morbidity e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months, ongoing infection as manifested by fever.
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test (serum or urine) at baseline. (Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential).
* Any prior chemotherapy or radiation for treatment of the patient's pancreatic tumor.
* Diagnosis for other invasive carcinomas (except basal cell carcinoma/squamous cell carcinoma of the skin) within the last five years. Carcinoma in-situ is allowed.
* Other serious uncontrolled medical conditions that the investigator feels might compromise study participation.
* Unwillingness to participate or inability to comply with the protocol for the duration of the study.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance or oral drug intake.
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment, without complete recovery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ryan, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Folfirinox-ARM A: Upon registration patients will be randomized to Arm A (FOLFIRINOX) or Arm B (Gemcitabine/nab-Paclitaxel
  * Treatment will be administered on an outpatient basis and will include intravenous administration of the FOLFIRINOX regimen on predetermined days.
  * After completion of FOLFIRINOX all patients without progressive disease will proceed with radiation therapy with the standard dose of capecitabine.
  * Between 2 and 4 weeks after radiation is complete, patients will proceed for surgical resection of pancreatic cancer
  FOLFIRINOX
  Radiation therapy
  Capecitabine
- Gemcitabine/Nab-Paclitaxel- Arm B: * Treatment will be administered on an outpatient basis. Upon registration patients will be randomized to Arm A (FOLFIRINOX) or Arm B (Gemcitabine/nab-Paclitaxel).
  * Intravenous administration of the Gemcitabine/Nab-paclitaxel regimen on predetermined days of each 28 day treatment cycle (unless a delay is mandated by toxicity criteria). A cycle of Gemcitabine/Nab-paclitaxel will constitute a 28 day treatment period.
  * After Gemcitabine/Nab-paclitaxel, all patients without progressive disease will proceed to radiation therapy with the standard dose of capecitabine
  * Between 2 and 4 weeks after radiation is complete, patients will proceed for surgical resection of pancreatic cancer
  Gemcitabine/nab-Paclitaxel
  Radiation therapy
  Capecitabine
Period: Overall Study
Arm/Group | Folfirinox-ARM A | Gemcitabine/Nab-Paclitaxel- Arm B
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Folfirinox-ARM A | Gemcitabine/Nab-Paclitaxel- Arm B | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Median (Full Range); unit: years] | 63.4 [49.4 to 68.3] | 71.9 [59.9 to 74.1] | 65.6 [49.4 to 74.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate at 18 Month
Description: Number of participants surviving after 18 months of study follow-up
Time Frame: 18 Month
Measure: Count of Participants; unit: Participants
Arm/Group | Folfirinox-ARM A | Gemcitabine/Nab-Paclitaxel- Arm B
Number analyzed (Participants) | 4 | 3
Participants | 2 | 3

2. Secondary Outcome: Pathologic Complete Response Rate (pCR).
Description: Number of patients achieving pathologic complete response at 18 months. Pathologic complete response is defined as the absence of residual invasive disease in the panaceas and in the regional lymph nodes.
Time Frame: 18 Months
Population: No Data available. Study terminated before any patients reached 18 months of follow-up. Patients were not able to be evaluated for response.
Arm/Group | Folfirinox-ARM A | Gemcitabine/Nab-Paclitaxel- Arm B
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

3. Secondary Outcome: Overall Survival Rate
Description: Overall survival rate at five years using Kaplan-Meier survival analysis
Time Frame: Baseline, 5 Years
Population: Study terminated before endpoint was reached, no data available
Arm/Group | Folfirinox-ARM A | Gemcitabine/Nab-Paclitaxel- Arm B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Number of Participants with Serious and Non-Serious Adverse Events from baseline to 28 days
Time Frame: Baseline, 28 Days
Measure: Number; unit: participants
Arm/Group | Folfirinox-ARM A | Gemcitabine/Nab-Paclitaxel- Arm B
Number analyzed (Participants) | 4 | 3
participants
  Serious Adverse Events | 0 | 2
  Other Adverse Events | 4 | 3

5. Secondary Outcome: Surgical Morbidity Rate
Description: Number of patients experiencing a specific surgery related morbidity
Time Frame: within 30 days of surgery
Population: Study ended prematurely, no results available
Arm/Group | Folfirinox-ARM A | Gemcitabine/Nab-Paclitaxel- Arm B
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

6. Secondary Outcome: 30-day Post-operative Mortality Rate
Description: Number of patients who died following surgery.
Time Frame: 30 Days
Population: Study ended prematurely, no results available
Arm/Group | Folfirinox-ARM A | Gemcitabine/Nab-Paclitaxel- Arm B
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

7. Secondary Outcome: Correlation of Biomarkers With PFS
Description: Analysis of the correlation between selected bio-markers and progression free survival.
Time Frame: 2 Years
Population: Data not available. Study was terminated before endpoint was able to be evaluated
Arm/Group | Folfirinox-ARM A | Gemcitabine/Nab-Paclitaxel- Arm B
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

8. Secondary Outcome: Rate of Pathologic Downstaging
Description: The number of participants achieving a reduction in the pathological staging of the primary cancer.
Time Frame: 2 Years
Population: Data not available. Study was terminated before endpoint was able to be evaluated
Arm/Group | Folfirinox-ARM A | Gemcitabine/Nab-Paclitaxel- Arm B
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

9. Secondary Outcome: Local Control Rate
Description: The number of participants achieving local control. The local control rate is defined as the number of participants achieving stable disease, partial response, or a complete response.
Time Frame: 2 Years
Population: Data not available. Study was terminated before endpoint was able to be evaluated
Arm/Group | Folfirinox-ARM A | Gemcitabine/Nab-Paclitaxel- Arm B
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Time Frame: Toxicity was assessed on day 1 of each cycle for the FOLFIRINOX arm and on Day 1, 8, 15 of each cycle for the Gem/Nab-P arm while being treated. Toxicity was assessed weekly during neoadjuvant radiation treatment and Capecitabine. Toxicity was planned to be assessed every 6 months during the first 3 years of post treatment follow-up.
Description: Toxicity was assessed with the use of physical exams, laboratory tests, and patient self reports.
Arm/Group | Folfirinox-ARM A | Gemcitabine/Nab-Paclitaxel- Arm B
All-Cause Mortality (participants affected / at risk) | 2/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Folfirinox-ARM A (N=4) | Gemcitabine/Nab-Paclitaxel- Arm B (N=3)
hypotension (Vascular disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Folfirinox-ARM A (N=4) | Gemcitabine/Nab-Paclitaxel- Arm B (N=3)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (7) | 2 (3)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (6) | 3 (4)
Fever (General disorders) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (6) | 2 (6)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2)
Weight loss (Investigations) | 2 (2) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No